CLINICAL TRIAL: NCT06917586
Title: Long Term Patient Outcomes and Product Durability of the Mosaic Mitral Valve Bioprosthesis in Patients Under 65
Brief Title: Mosaic Mitral Valve: Long-Term Outcomes in Patients Under 65
Acronym: MMV
Status: Recruiting | Type: Observational
Sponsor: Michael Moront (Other)
Responsible Party: Sponsor-Investigator, Michael Moront, Doctor Of Medicine, ProMedica Health System
Organization: ProMedica Health System (Other)
Other Study IDs: IRB# 24-129; ERP-2024-13849 (Other Grant/Funding Number: Medtronic, Inc)
Record Dates: First submitted 2024-12-16; First posted 2025-04-08 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-03

CONDITIONS: Valve Disease, Heart; Valve Replacement; Valve Regurgitation, Mitral; Valve Heart Stenosis
Keywords: Mitral Valve; Bioprosthetic; Mosaic; Valvulopathy
MeSH Terms: conditions — Heart Valve Diseases; Mitral Valve Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Mitral Valve Replacement: Patients who have undergone mitral valve replacement at ProMedica Hospital using the mosaic bioprosthesis and were under the age of 65.

SUMMARY:
The safety and efficacy of the Mosaic bioprosthetic heart valves for cardiac valve replacement in the aortic position has been well documented throughout the literature. However, few studies assessing structural valve deficiency, patient outcomes and overall product performance in patients under the age of 65 exists for the Mosaic mitral valve bioprosthetic. This study aims to assess valve efficacy, stability, and post operative outcomes in patients who have received the Mosaic mitral valve prothesis at ProMedica Toledo Hospital and were under the age of 65.

DETAILED DESCRIPTION:
Background:

Within the U.S., the prevalence of valvular heart disease is estimated at 2.5% with an abrupt increase after the age of 65 years, predominantly due to degenerative etiologies. In patients with significant valve insufficiency or stenosis where repair or reconstruction is not feasible, valve replacement is the most offered solution. The two types of heart valves offered to patients include mechanical or bioprosthetic. The major advantage of bioprosthetic heart valves in comparison to mechanical valves is the lack of post-operative anticoagulant therapy. However, the major disadvantage of bioprosthetic heart valves lie in their reduced durability compared to mechanical valves, with reoperation rates of ~10% at 10 years and up to 30% at 15 years.

The use of porcine bioprosthetic heart valves for cardiac valve replacement first appeared in the late 1960s and have been widely used since due to the avoidance of anticoagulant therapy. One of the major drawbacks associated with bioprosthetic valves is structural valve deterioration (SVD) which can lead to reduced valve durability, necessitating reoperation. The causes of SVD are poorly understood, however, it is thought to result from the accumulation of calcium and lipids on the valve surface. The Medtronic Mosaic mitral bioprosthetic valve is a 3rd-generation, stented porcine heart valve that was originally approved for clinical use in the U.S. in 2000. These valves are treated with a 0.2% glutaraldehyde solution stabilizing the tissue by cross-linking free lysine residues. In addition, the valve is treated with alpha-amino oleic acid (AOATM) which has been shown to mitigate leaflet calcification in animal studies. Long term clinical safety and efficacy of the Mosaic valve in the aortic position is well documented throughout the literature however, few studies exist detailing performance in the mitral position. Moreover, even fewer studies exist detailing overall valve survival in patients under 65 due to the more common recommendation of the use of mechanical valve replacement in this population. The purpose of this study is to examine long-term outcomes in patients who have received the Mosaic mitral valve bioprosthetic and were under the age of 65 at placement.

Significance:

The investigation of the Medtronic mosaic heart valve in the mitral position will allow for a better assessment of product performance and its impact on patient outcomes. Results can inform physicians on the longevity of the product when used in the mitral position allowing for more accurate prediction of replacement time. In addition, the results may provide further information to the safety and efficacy of placement in the mitral position in patients under the age of 65, a population in which mechanical valves are more prevalent.

ELIGIBILITY:
Inclusion Criteria:

* Received the Mosaic Mitral Valve Bioprosthetic at ProMedica Toledo Hospital
* Under the age of 65

Exclusion Criteria:

* Over the age of 65
* Under the age of 18
* Surgery performed at institutions outside of ProMedica Toledo Hospital

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population will include patients who received the mosaic mitral valve bioprosthetic and were between 18-65 years of age at the time of surgery.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Mortality | From January 2001 to December 2025
  Mortality in patients who were under the age of 65 when receiving the mosaic mitral valve bioprosthetic at ProMedica hospital. Patient records will be reviewed to determine mortality rate of patients who were under 65 years of age when receiving the mosaic mitral valve bioprosthetic.
Morbidity | January 2001 - December 2025
  Post operative morbidity rate for a series of outcomes will be assessed in patients who received the Mosaic mitral valve bioprosthetic over time.

SECONDARY OUTCOMES:
Valve Stability | From January 2001 to December 2025
  Assess valve stability in patients who received a mosaic mitral valve bioprosthetic at ProMedica Toledo Hospital. Valve stability will be assessed by reviewing post operative echocardiographic data.
Freedom of Re-operation | January 2001 - December 2025
  A survival analysis for freedom of reoperation will be assessed for patients who were under 65 at the time of mitral valve replacement.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Moront, MD, Principal Investigator — ProMedica Health System
Locations (1):
- ProMedica Toledo Hospital, Toledo, Ohio, United States

IPD SHARING:
Plan to Share IPD: No